CLINICAL TRIAL: NCT05745363
Title: Phase Ib Clinical Trial to Evaluate the Efficacy and Safety of AL2846 Capsule in Iodine-resistant Differentiated Thyroid Cancer With Previous TKI Treatment Failure
Brief Title: Clinical Study of AL2846 Capsule in the Treatment of Differentiated Thyroid Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL2846-Ib-02
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Differentiated Thyroid Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AL2846 capsule (Experimental): AL2846 capsules monotherapy, 28 days as a treatment cycle.
  Interventions: Drug: AL2846 capsule

INTERVENTIONS:
Drug: AL2846 capsule — AL2846 is a multi-target tyrosine kinase inhibitor

SUMMARY:
This is a Phase Ib clinical trial to evaluate the efficacy and safety of AL2846 capsule in iodine-refractory differentiated thyroid cancer that has failed previous TKI treatment. The trial is planned to enroll 20 subjects. The trial is a single-arm, multi-center, open label clinical study. Objective response rate (ORR) is the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18~80 years old (when signing the informed consent form), regardless of gender;
* Differentiated thyroid carcinoma (DTC) confirmed by histopathology or cytology;
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumours (RECIST 1.1);
* Disease progression occurs after receiving at least one (but not more than two) Vascular Endothelial Growth Factor Receptor (VEGFR) targeted therapy in the past;
* Iodine refractory patients can be defined as iodine refractory if they meet one of the following conditions:

  1. The lesions showed no iodine uptake on the whole body imaging after 131I treatment, and could not benefit from the follow-up 131I treatment (it must be confirmed by the endocrinologist or nuclear medicine physician. If there are too many residual thyroid, it may affect the iodine uptake of the metastatic lesions, which can be evaluated when the thyroid is removed and treated again);
  2. The lesions that originally took iodine gradually lost the ability to take iodine after 131I treatment;
  3. Some lesions in the same patient take iodine, while some lesions do not take iodine, and there is no biochemical remission;
  4. The focus takes iodine, but the disease progresses within 12 months (confirmed by imaging);
  5. The cumulative dosage of 131I ≥ 600mCi or 22GBq, but the disease did not alleviate (confirmed by imaging).
* There was evidence of imaging progress within 14 months before the knowledge;
* Thyroid Stimulating Hormone (TSH) ≤ 0.5mIU/L under the treatment of TSH inhibitor;
* Eastern Cooperative Oncology Group (ECOG) score: 0-1;
* Estimated survival time ≥ 12 weeks;
* Normal function of main organs
* HBsAg positive patients must meet the requirements of Hepatitis B Virus (HBV) DNA compliance or receive anti-HBV treatment at least one week before the start of the study, and the virus index is reduced by more than 10 times. At the same time, the patients are willing to receive anti-HBV treatment throughout the whole study period; The patients with hepatitis C antibody positive and Hepatitis B Virus (HCV) RNA quantitative positive should complete antiviral treatment at least 1 month before starting the study; 12) The serum Human Chorionic Gonadotropin (HCG) test of female patients of childbearing age must be negative within 7 days before study enrollment and must be non-lactating; The patient should agree to use contraception during the study period and within 6 months after the end of the study period; 13) The patient voluntarily joined the study and signed the informed consent form, with good compliance.

Exclusion Criteria:

* Combined with the following diseases or medical history:

  1. Have undifferentiated thyroid cancer or medullary thyroid cancer;
  2. Known thyroid cancer with Rearranged during Transfection (RET) fusion positive;
  3. Other malignant tumors have occurred or are present at the same time within<3 years before the first administration. The following two cases can be included in the group: other malignant tumors treated by single surgery have achieved R0 resection without recurrence and metastasis; Cured cervical carcinoma in situ, skin basal cell carcinoma and superficial bladder tumor [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
  4. CTCAE5.0 ≥ grade 2 therapeutic toxicity caused by any previous treatment that has not been completely relieved, excluding hair loss;
  5. Inability to tolerate multiple factors affecting oral medication due to any reason;
  6. Major surgical treatment or obvious traumatic injury (excluding puncture for diagnosis, endoscopic biopsy, etc.) was received within 4 weeks before the first administration;
  7. Wounds or fractures that have not been cured for a long time;
  8. Arterial/venous thrombosis events occurred within 6 months before the first administration, such as cerebrovascular accident, deep venous thrombosis and pulmonary embolism;
  9. Those who have a history of abuse of psychotropic substances and are unable to quit or have mental disorders;
  10. Subjects with any severe and/or uncontrollable disease, including:

      1. Poor blood pressure control (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg);
      2. Patients with ≥ grade 2 myocardial ischemia or myocardial infarction, arrhythmia (including male corrected QT interval ≥ 450ms, female corrected QT interval ≥ 470ms) and ≥ grade 2 congestive heart failure (New York Heart Association (NYHA) classification);
      3. Active or uncontrolled serious infection (≥ CTCAE grade 2);
      4. Decompensated stage of liver cirrhosis;
      5. Renal failure requiring hemodialysis or peritoneal dialysis;
      6. Have a history of immunodeficiency, including HIV-positive or other acquired and congenital immunodeficiency diseases, have received allogeneic hematopoietic stem cell transplantation, solid organ transplantation or have received autologous hematopoietic stem cell transplantation within 12 weeks before the first administration;
      7. Poor control of diabetes (FBG>10mmol/L);
      8. Those who have epilepsy and need treatment;
* Tumor related symptoms and treatment:

  1. Have received surgery, chemotherapy, radiotherapy (brain radiotherapy for 2 weeks) or other anti-cancer therapy within 4 weeks before the first administration;
  2. Participated in clinical trials of other anti-tumor drugs within 4 weeks before the first administration;
  3. Any type of small-molecule kinase inhibitor has been accepted within 2 weeks before the first administration;
  4. Within 2 weeks before the first administration, he has received the treatment of traditional Chinese medicine with anti-tumor indications specified in the drug instructions approved by China National Medical Products Administration;
  5. Uncontrolled pleural effusion, pericardial effusion or ascites that still need repeated drainage (judged by the investigators);
* Others:

  1. Vaccination history of live attenuated vaccine within 4 weeks before the first administration or live attenuated vaccine is planned during the study period;
  2. Allergic to known ingredients of AL2846 capsule;
  3. According to the judgment of the researcher, there are patients with concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or those who think there are other reasons that are not suitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | From baseline up to 12 months.
  ORR is defined as the percentage of participants with complete remission (CR) and partial remission (PR) based on investigator records.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From baseline up to 12 months.
  PFS is defined as the time from randomization to the first recorded progressive disease (PD) or death from any cause.
Disease control rate (DCR) | From baseline up to 12 months.
  DCR is defined as the percentage of patients who have achieved complete response, partial response and stable disease.
Duration of remission (DoR) | From baseline up to 12 months.
  The time from the start of the first evaluation of the tumor as CR or PR to the first assessment as PD or death from any cause.
Overall survival (OS) | From baseline to death event.
  Time from the first administration to death due to any cause.
Occurrence of all adverse events (AEs) | From baseline to 28 days after the last dose or start of a new antineoplastic therapy (whichever comes first).
  Adverse events are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Affiliated Hospital Of Guilin Medical University, Guilin, Guangxi
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Yunnan Cancer Hospital, Kunming, Yunnan